CLINICAL TRIAL: NCT03666481
Title: Psychosocial Effects of a Motivational Physical Activity Program in Bariatric Patients
Brief Title: Physical Activity in Bariatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Collaborators: Fundacion MAPFRE (Other); Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, David González-Cutre Coll, PhD, Universidad Miguel Hernandez de Elche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UEM2.11X
Record Dates: First submitted 2018-07-13; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate
Keywords: Sleeve gastrectomy; Accelerometer; Exercise; Self-determination theory; Morbid obesity
MeSH Terms: conditions — Obesity, Morbid; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MPAI group (Experimental): Patients in this group participated in a 6-months Motivational Physical Activity Intervention (MPAI) to explore its effects on different variables related to PA levels and psychosocial aspects of life of bariatric patients. Concretely, the fundamental goals of the MPAI group were three: to increase the self-determined forms of motivation of the patients towards exercise or reduce those related to non-self-determined motivation; to improve post-operative levels of PA with respect to pre-operative levels, and; transfer the benefits of the intervention on different variables related to the perceived health-related quality of life.
  Interventions: Behavioral: Motivational Physical Activity Intervention (MPAI)
- Control group (No Intervention): Patients in this group did not participate in any intervention, but the same measurements were made in them as in the MPAI group in the same temporal spaces.

INTERVENTIONS:
Behavioral: Motivational Physical Activity Intervention (MPAI) — MPAI was carried out during 6 consecutive months. The sessions were directed by sport sciences professionals, who were trained in the application of motivational strategies based on self-determination theory.
  The frequency of training, as well as the duration of the sessions, was increasing throughout the 6 months. The contents of the sessions could be directed in two ways: sessions with activities to develop cardiorespiratory fitness and muscular strength, and playful sessions to enhance psychosocial aspects. Nevertheless, motivational strategies were implemented in both types of sessions.
  Arms: MPAI group

SUMMARY:
The aim of the current study was to explore the effect of a 6-months motivational physical activity intervention (MPAI) on different psychosocial variables (e.g. motivation, health-related quality of life, self-esteem, etc.) and on the physical activity levels of bariatric surgery patients. Comparing with a control group (CG), we tested the differences obtained on these variables between before surgery and just after the MPAI (7-months after surgery). Additionally, we explored the (possible) prolonged effects of the intervention by doing re-tests 13, 25 and 37- months after surgery.

DETAILED DESCRIPTION:
Participants were recruited from a Spanish hospital between November 2011 and May 2013. Through their pre-operative visit to the clinical psychologist, patients were asked if they wanted to participate in a follow-up intervention to measure their physical activity (PA) levels and various psychological variables related to exercise. Participants who showed interest after this interview were subsequently contacted by phone to arrange a baseline visit to the sport research center, during which they were informed about the aims and procedure of the study, provided written consent, and completed questionnaires to assess different variables related to psychosocial aspects. Moreover, participants were asked to wear an accelerometer at their right hip for one week, warning them to take it off just to sleep, shower, or to perform activities that could damage the device (e.g. swimming). When they returned, they were assigned to a motivational PA intervention (MPAI) or control (CG) group.

At post-intervention measurements, patients again completed all questionnaires and wore an accelerometer during another week.

Regarding the MPAI, it was carried out during 6 consecutive months and took place in a public fitness center. The sessions were directed by exercise and sport sciences professionals (Degree in sport sciences, Master's degree in PA and health), who were trained in the application of motivational strategies based on self-determination theory (SDT). According with the postulates of SDT, these motivational strategies would help to enhance the satisfaction of basic psychological needs that are necessary for optimal development and functioning, such as competence, autonomy, relatedness and novelty. So, in the context of exercise, intrinsic forms of motivation will appear in people if basic psychological needs are satisfied, which will lead to positive consequences related to enjoyment, adherence, and positive attitudes towards PA.

ELIGIBILITY:
Inclusion Criteria:

* To have a BMI greater than 40kg/m2 or greater than 35kg/m2 with an associated comorbidity.
* To have experienced previous failed obesity treatments with restrictive-caloric diets and medications.
* To have followed endocrinology and nutritional monitoring, accomplishing the therapeutic instructions properly.
* To have no medical, psychological or social contraindications.
* To have the consent of the clinical psychiatrist and the surgeon and ensure their willingness to attend the programme.

Exclusion Criteria:

* To participate in another physical activity or weight loss program
* Not ensuring full availability to attend the program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11-16 (Actual); Primary Completion 2015-05-15 (Actual); Study Completion 2015-10-15 (Actual)

PRIMARY OUTCOMES:
Changes in objective physical activity levels. | From before surgery to after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  GT3X accelerometers were used to measure changes in objective physical activity levels. Participants were asked to wear the accelerometer at the right hip during 7 consecutive days, considering minimal wear time required to estimate PA a total of ≥ 3 days with at least ≥ 10 hours wear time per day at all measurements. Vector magnitude activity counts, calculated as the square root of the sum of the vertical, medio-lateral and antero-posterior axes was used according to previous studies performed with this population. Non-wear time was defined as 60 min of consecutive zeros, allowing for 2 min of non-zero interruptions. Time spent sedentary was defined as all minutes showing less than 100 counts per minute (cpm), light PA as 101-3027 cpm, moderate PA as 3028-8564 cpm and vigorous PA as number of minutes showing more than 8565 cpm.
Changes in self-reported physical activity levels. | From before surgery to after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  The Spanish version of the Seven-Day Physical Activity Recall (7-Day PAR) questionnaire was used to assess changes in self-reported levels of physical activity. Participants must indicate the minutes dedicated every day of the week to physical activity, distinguishing between different intensities: moderate ("activities that feel like walking at a normal pace"), hard ("activities that are not as intense or hard as running, but requiring more effort than moderate activity"), and very hard ("activities that feel like running"). The questionnaire also collects information about the participants' daily hours of sleep. The questionnaire protocol allowed us to calculate the total minutes of daily light activity by subtracting the time dedicated to sleeping and to moderate, hard, and very hard physical activity from the total minutes of the day.
Changes in health-related quality of life. | From before surgery to after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  The Spanish version of the Medical Outcomes Study Short-Form 36 Health Status Survey (SF-36) was used to measure patients' quality of life in physical and mental domains. This questionnaire measures eight domains of functioning and obtains a physical component score (PCS) and a mental component score (MCS). So, PCS is composed by four domains, such as physical functioning, role-limitations because of physical problems, bodily pain, and general health. MCS, on the other hand, is composed by social functioning, role-limitations because of emotional problems, vitality, and mental health. Both PCS and MCS are obtained by calculating the average of their respective factors. Scores ranged from 0 (worst possible level of functioning) to 100 (best possible level of functioning) for all variables. The scores were standardized according to the normative values for the Spanish context.
Changes in physical activity motivation. | From before surgery to after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  The Spanish version of the Behavioural Regulation in Exercise Questionnaire-3 (BREQ-3) was used to changes in physical activity motivation. The BREQ-3 includes 23 items, rated on a 4-point Likert-scale, from 0 ("not true of me") to 4 ("very true of me") that assess motivation types based on continuum conception of extrinsic and intrinsic motivation established by self-determination theory. Non self-determined types of motivation would be represented by amotivation, external regulation and introjected regulation, while self-determined forms of motivation would be composed by identified regulation, integrated regulation and intrinsic regulation. The means of each subscale are calculated separately to check the scores of each type of motivation.
Changes in patients' needs satisfaction in their general life. | From before surgery to after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  The Spanish version of the Basic Needs Satisfaction in General Scale (BNSG-S) was used to measure patients' needs satisfaction in their general life. The BNSG-S includes 21 items, rated on a 7-point Likert-scale, from 1 ("not true of me") to 7 ("very true of me") that assess the basic psychological needs of autonomy, competence and relatedness. We also measure satisfaction of the need for novelty. The means of each subscale are calculated separately to check the scores of each need. In this way, lower scores indicate lower satisfaction of basic psychological needs, and vice versa.
Measurement of the patients' needs satisfaction in exercise settings. | After the MPAI (7-months post-surgery)
  The Spanish version of the Basic Psychological Needs in Exercise Scale (BPNES) was used to measure patients' needs satisfaction in exercise settings. The BPNES includes 12 items, rated on a 5-point Likert-scale, from 1 ("totally disagree") to 5 ("totally agree") that assess the basic psychological needs of autonomy, competence and relatedness in exercise settings. The means of each subscale are calculated separately to check the scores of each need. In this way, lower scores indicate lower satisfaction of basic psychological needs, and vice versa.
Measurement of the patients' perception of autonomy support provided by instructors. | After the MPAI (7-months post-surgery)
  The Spanish version of the Perceived Autonomy Support Scale for Exercise Settings (PASSES) was used as a tool to measure the perception of autonomy support provided by instructors. The PASSES includes 12 items, rated on a 7-point Likert-scale, from 1 ("totally disagree") to 7 ("totally agree") that assess the autonomy support perceived by patients when they participated in the MPAI. Therefore, scores close to 7 refer to a positive perception of autonomy support, while scores close to 1 refer to the fact that patients hardly felt that autonomy support.
Changes in patients' concerns about their body shape. | From before surgery to after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  The Spanish version of the Body Shape Questionnaire (BSQ) was used to measure patients' concerns about their body shape. The BSQ includes 34 items, rated on a 6-point Likert-scale, from 1 ("never") to 6 ("always"). The total score is obtained by summing the scores of each of the 34 items. Higher scores express greater dissatisfaction with the body, and vice versa.
Changes in patients' self-esteem. | From before surgery to after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  The Spanish version of the Rosenberg Self-Esteem Scale (RSES) was used as an instrument for evaluating changes in participants' self-esteem. This tool is a 10-item scale which measures global self-worth by calculating both positive and negative feelings about the self. All items are answered using a 4-point Likert scale format ranging from "strongly agree" to "strongly disagree". The total score is obtained by summing all 10 items. Higher scores indicate higher self-esteem.
Changes in patients' satisfaction with life. | From before surgery to after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  The Spanish version of the Satisfaction with Life Scale (SWLS) was used to measure patients' satisfaction with life. The SWLS includes 5 items, rated on a 5-point Likert-scale, from 1 ("totally disagree") to 5 ("totally agree"). The total score is obtained by summing the score of all items and dividing it by 5 (average of the items), in such a way that higher scores express greater satisfaction with life and vice versa.
Changes in types of motivation in health, leisure and relation activities. | From before surgery to after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  The Spanish version of the Elderly Motivation Scale (EMS) was used to measure different types of motivation in three life domains (health, leisure and relation activities). Concretely, we used the EMS to measure changes in intrinsic motivation, self-determined extrinsic motivation, non self-determined extrinsic motivation and amotivation in health, leisure and relation activities. The EMS includes 9 questions (3 questions by life domain). Each question has 4 items, rated on a 7-point Likert-scale from 1 ("Absolutely disagree") to 7 ("Absolutely agree"), that measure intrinsic motivation, amotivation, non self-determined extrinsic motivation and self-determined extrinsic motivation, respectively. Thus, the EMS has a total of 12 items per life domain and a grand of 36 items for the whole scale. The total score for each life domain is obtained by summing the score of the items related with each type of motivation and dividing it by 3 (average of the items).

SECONDARY OUTCOMES:
Sex | At baseline (before surgery)
  The variable "sex" was collected as part of the sociodemographical variables.
Age | At baseline (before surgery)
  The variable "age" was collected as part of the sociodemographical variables.
Height | At baseline (before surgery)
  The variable "height" was collected as part of the sociodemographical variables.
Weight | Before surgery, after the MPAI (7-months post-surgery) and 13, 25 and 37- months post-surgery.
  The variable "weight" was collected as part of the sociodemographical variables.
Educational level | At baseline (before surgery)
  The variable "educational level" was collected as part of the sociodemographical variables.
Race/ethnicity | At baseline (before surgery)
  The variable "race/ethnicity" was collected as part of the sociodemographical variables.
Marital status | At baseline (before surgery)
  The variable "marital status" was collected as part of the sociodemographical variables.
Addictive behaviours | At baseline (before surgery)
  The variable "addictive behaviours" was collected as part of the sociodemographical variables.

CONTACTS AND LOCATIONS:
Overall Officials: David González-Cutre, PhD, Principal Investigator — Sport Research Center. Miguel Hernández University of Elche.
Locations (1):
- Sport Research Center. Miguel Hernández University of Elche., Elche, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bond DS, Vithiananthan S, Thomas JG, Trautvetter J, Unick JL, Jakicic JM, Pohl D, Ryder BA, Roye GD, Sax HC, Wing RR. Bari-Active: a randomized controlled trial of a preoperative intervention to increase physical activity in bariatric surgery patients. Surg Obes Relat Dis. 2015 Jan-Feb;11(1):169-77. doi: 10.1016/j.soard.2014.07.010. Epub 2014 Jul 30. PMID 25304832
- [Result] Bond DS, Graham Thomas J, Vithiananthan S, Webster J, Unick J, Ryder BA, Pohl D. Changes in enjoyment, self-efficacy, and motivation during a randomized trial to promote habitual physical activity adoption in bariatric surgery patients. Surg Obes Relat Dis. 2016 Jun;12(5):1072-1079. doi: 10.1016/j.soard.2016.02.009. Epub 2016 Feb 17. PMID 27246138
- [Result] Berglind D, Willmer M, Eriksson U, Thorell A, Sundbom M, Udden J, Raoof M, Hedberg J, Tynelius P, Naslund E, Rasmussen F. Longitudinal assessment of physical activity in women undergoing Roux-en-Y gastric bypass. Obes Surg. 2015 Jan;25(1):119-25. doi: 10.1007/s11695-014-1331-x. PMID 24934315
- [Result] Berglind D, Willmer M, Tynelius P, Ghaderi A, Naslund E, Rasmussen F. Accelerometer-Measured Versus Self-Reported Physical Activity Levels and Sedentary Behavior in Women Before and 9 Months After Roux-en-Y Gastric Bypass. Obes Surg. 2016 Jul;26(7):1463-70. doi: 10.1007/s11695-015-1971-5. PMID 26613756